CLINICAL TRIAL: NCT00982709
Title: The Effects of Treadmill Versus Agility Training in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Fay B. Horak, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4402
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Exercise; Parkinson's Disease
MeSH Terms: conditions — Motor Activity; Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Types (Active Comparator): comparing two different exercise programs for PD
  Interventions: Behavioral: Aerobic vs. Agility Training

INTERVENTIONS:
Behavioral: Aerobic vs. Agility Training — High Intensity 4x's per week for 4 weeks with a physical therapist.
  Other Names: agility, treadmill

SUMMARY:
Aim:

To determine the Responsiveness of the iMOBILITY in response to intensive physical therapy exercise programs. (Is it sensitive to change?) Although exercise is thought to be the most effective intervention for balance and gait in PD (compared to dopaminergic medication or DBS surgery), the best exercise program for mobility in PD is unknown. The iMOBILITY will be used to quantify balance and gait performance before and after two PT-supervised, intensive, exercise programs, expected to improve balance and gait. The first program is a published Treadmill training program and the second is the investigators new Agility training program with sensorimotor progressions, targeted at specific impairments that underlie the abnormalities of balance and gait in PD (developed for the Kinetics Foundation). This pilot clinical trial will randomize 40 PD subjects into the two exercise programs at OHSU in preparation for a larger clinical trial to determine the most effective exercise for mobility disability in PD. The effects of exercise will be compared with no treatment during a 5-week delay prior to start of exercise.

This trial will also determine the relative responsiveness (compared to traditional clinical scales) of the iMOBILITY for testing the hypothesis that intensive exercise can improve mobility in PD. We will use existing instruments (Berg Balance Scale, BEST of dynamic balance, UPDRS, PDQ-39, 5 times sit-to-stand time and the Functional Performance Battery) to show there is a difference between the exercise groups. Superior responsiveness of the iMOBILITY system will be determined by larger differences with exercise intervention with the iMOBILITY system than with traditional clinical measures of mobility in PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic PD

Exclusion Criteria:

* Other neurological conditions, artificial joints

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Dynamic Posturography | pre and post intervention

SECONDARY OUTCOMES:
UPDRS | pre and post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886